CLINICAL TRIAL: NCT02262065
Title: Individual Risk Factors for Enhanced Inflammation to Arthroplasty Wear Particles: Analysis of Cytokine Polymorphisms and in Vitro Cytokine Production to Wear Particles (Ceramic, Metal, XPE)
Brief Title: Risk Factors for Enhanced Inflammation to Arthroplasty Wear Particles: Analysis of Cytokine Production and Polymorphisms
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Technical University of Munich (Other); University of Rostock (Other)
Responsible Party: Principal Investigator, Peter Thomas, Prof. Dr., Ludwig-Maximilians - University of Munich
Other Study IDs: 230-12
Record Dates: First submitted 2013-12-23; First posted 2014-10-10 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Allergy; Implants
Keywords: implant; allergy; particle; cytokine
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples of 20 patients (subgroup analysis)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients with suspected arthroplasty intolerance
- Controls: Patients with well tolerated arthroplasties

SUMMARY:
Assessment of cytokine polymorphisms in 100 patients with aseptic complications to arthroplasty as compared to 100 symptom-free arthroplasty patients.

In selected patients additional in-vitro cytokine release assay with peripheral blood mononuclear cells (PBMC) stimulated with different wear particles.

DETAILED DESCRIPTION:
A cytokine polymorphism analysis in 100 individuals with aseptic implant intolerance reaction (patients of the implant allergy special ambulance) and in 100 asymptomatic patients with implanted endoprostheses will be done. Furthermore, supplementary clinical data (such as type of implant, hospital stay, discomfort), questionnaire-based history and a clinical score (WOMAC score) are recorded. In the subgroup analysis in 10 patients of implant patients with complaints with special found cytokine polymorphisms and 10 implant patients without problems the cytokine response to particles in vitro will assessed.

Test parameters:

1. total collective:

   the DNA of cryopreserved blood sample will be isolated. By polymerase chain reaction, four different known polymorphisms will be analyzed, three IL-1B genes (IL-1B-3954 IL-1B-31, and IL-1B-511), and a IL-1ß receptor antagonist gene (IL -1-RN, intron 2 VNTR). Molecular analysis includes DNA isolation, polymerase chain reactions (PCR) and gel electrophoresis.
2. Subgroup analysis:

Peripheral blood cells will be isolated from 10 implant patients with complications and 10 symptom-free persons and stimulated in cell culture with control stimuli, the IL-1ß-inducer lipopolysaccharide (LPS) and ceramic particles (BIOLOX delta)*, CoCrMo particles and XPE-particles** cultured separately or in combination. The secretion of IL-1ß and selected proinflammatory cytokines will be measured. The methods include cell isolation by density centrifugation and analysis of cell culture supernatants by a multiplex cytokine measurement assay by flow cytometry.

* Supplied CeramTec

** Generated and processed by the Working Group of the cooperation partner Prof. R. Bader (University Hospital Rostock) in special carrier system for cell culture stimulation approach

ELIGIBILITY:
Inclusion Criteria:

* arthroplasty
* over 18 years
* no infection

Exclusion Criteria:

* inability to consent
* malposition
* infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with arthroplasty:
  A) without symptoms B) with aseptic complications
Sampling Method: Non-Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2012-07; Primary Completion 2018-01 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Polymorphism frequency | 2 years
  Frequency of 4 different cytokine polymorphisms will be assessed in the 2 study groups.

SECONDARY OUTCOMES:
Cytokine production | 1 year
  Subgroup analysis: In vitro cytokine production of 20 patients with special polymorphism constellation will be analyzed after stimulation with particles.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Thomas, Prof. Dr., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Ludwig-Maximilians-University Munich, Dept. of Dermatology, Munich, Bavaria, Germany